CLINICAL TRIAL: NCT04448457
Title: Sufentanil Sublingual Tablet System For Management Of Postoperative Pain In Enhanced Recovery After Surgery Pathway For Total Knee Arthroplasty: A Randomized Controlled Study
Brief Title: Sufentanil Sublingual Tablet System for Postoperative Pain Management After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Tivoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2017/348
Record Dates: First submitted 2020-06-24; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Postoperative Pain
Keywords: SSTS; Oxycodone; Enhanced recovery after surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Sufentanil; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSTS group (Experimental): Patients received sufentanil nanotab patient controlled analgesia (PCA) system (Zalviso) 15 mcg with 20 min of lockout interval during 48 hours postoperatively
  Interventions: Drug: Sufentanil Sublingual Tablet
- Oxycodone group (Active Comparator): Patients received oxycodone extended-release tablet (OxyContin) 10 mg every 12 hours systematically plus Oxycodone 5 mg every 6 hours if numeric rating scale is above 3 during the 48 hours postoperatively
  Interventions: Drug: Oxycodone oral tablet and oxycodone extended-release oral tablet

INTERVENTIONS:
Drug: Sufentanil Sublingual Tablet — 15 mcg with lockout interval of 20 min
  Other Names: Zalviso
  Arms: SSTS group
Drug: Oxycodone oral tablet and oxycodone extended-release oral tablet — Oxycodone hydrochloride 5 mg and Oxycodone extended-release 10 mg
  Other Names: OxyNorm; OxyContin
  Arms: Oxycodone group

SUMMARY:
The aim of this study is to assess the effectiveness of Sublingual Sufentanil Tablets System (SSTS, Zalviso ®) to control postoperative pain after total knee arthroplasty in the context of early rehabilitation program.

SSTS is a novel patient controlled analgesia system wich does not require intravenous access, potentially improving pain control and promoting mobilization.

SSTS will be randomly compared to nurse-driven oral Oxycodone.

DETAILED DESCRIPTION:
Even with multimodal analgesia (combining local anesthetic infiltration, corticosteroids, non-steroidal anti-inflammatory drugs and acetaminophen), total knee arthroplasty is associated with acute moderate-to-severe postoperative pain requiring opioids treatment. We compare the efficacy of SSTS and oral Oxycodone in this context.

After written informed consent, patients will be randomly assigned postoperatively to SSTS or Oral oxycodone group at a ratio 1:1. Pain scores, mobilization and patient satisfaction will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years)
* Scheduled for unilateral total knee arthroplasty under spinal anesthesia
* American Society of Anesthesiologists (ASA) class 1-3

Exclusion Criteria:

* Contraindication to medication used in our multimodal analgesia protocol (solumedrol, celecoxib, acetaminophen, ropivacaine)
* Allergy to study medications
* History of addiction or preoperative chronic use of opioids
* Unicompartmental or revision knee replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score assessed at 24 hours | 24 hours after surgery
  A numerical pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain at rest and dynamically 24 hours after surgery

SECONDARY OUTCOMES:
Postoperative pain scores assessed over 48 hours | 2 hours, 6 hours, 12 hours, 18 hours, 24 hours, 30 hours, 36 hours, 42 hours, 48 hours after surgery
  A numerical pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain at rest and dynamically
Time to first mobilization | 2 hours, 6 hours, 12 hours, 18 hours, 24 hours, 30 hours, 36 hours, 42 hours, 48 hours after surgery
  Successful mobilization with or without aid assessed at specific timepoints
Patient satisfaction | At completion of the study period of 48 hours
  Satisfaction for the method of pain control assessed using Patient Global Assessment (PGA) of the method of pain control questionnaire at the completion of the 48h study period which consist on a 4-point categorical scale, where 1 = poor, 2 = fair, 3 = good, and 4 = excellent.

OTHER OUTCOMES:
Incidence of nausea and vomiting | At completion of the study period of 48 hours
  Percentage of patients who experienced nausea or vomiting during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Noel, MD, Principal Investigator — Centre Hospitalier Universitaire de Tivoli
Locations (1):
- Chu Tivoli, La Louvière, Belgium

REFERENCES:
- [Derived] Noel E, Miglionico L, Leclercq M, Jennart H, Fils JF, Van Rompaey N. Sufentanil sublingual tablet system versus oral oxycodone for management of postoperative pain in enhanced recovery after surgery pathway for total knee arthroplasty: a randomized controlled study. J Exp Orthop. 2020 Nov 20;7(1):92. doi: 10.1186/s40634-020-00306-x. PMID 33216238